CLINICAL TRIAL: NCT01192386
Title: Eosinophil Markers and Development of Disease in Allergic Rhinitis. A 15-year Follow-up of Patients With Grass Pollen Induced Hayfever.
Brief Title: Eosinophil Markers and Development of Disease in Allergic Rhinitis
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Ass. professor Lars Peter Nielsen, Department of Respiratory Research, Aarhus University Hospital
Other Study IDs: RHINO2010
Record Dates: First submitted 2010-08-30; First posted 2010-09-01 (Estimated); Last update posted 2010-09-01 (Estimated); Status verified 2010-08

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
Inflammatory proteins from eosinophil granulocytes in blood from patients with seasonal allergic hayfever have been shown to predict development of asthma at a six-year follow-up. This study is a 15-year follow-up of the same patients to verify earlier results and study disease development.

DETAILED DESCRIPTION:
The study consists of a single visit at which patients fill in a questionnaire on actual hayfever and asthma symptoms as well as current treatment. Blood samples and nasal lavages are drawn and analysed for eosinophils as well as eosinophil cationic protein and tryptase. Spirometry is performed.

If patients use drugs which can interfere with results, ie. corticosteroids or beta-agonists, biochemistry and/or spirometry are omitted.

ELIGIBILITY:
Inclusion Criteria:

* Participant in earlier study (1995)

Exclusion Criteria:

* Treatment with any kind of corticosteroid within two months will exclude from study of inflammatory parameters

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Follow-up on participants in Allergic Rhinitis study 1995.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2010-05; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Asthma morbidity | Single measurement - May 2010
  Patients are asked whether they have experienced asthmatic symptoms or have been disgnosed with asthma within the latest 15 years

SECONDARY OUTCOMES:
Rhinitis morbidity | Single measurement - May 2010
  Patients are asked for current hayfever symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Lars Peter Nielsen, MD, Principal Investigator — Department of Respiratory Research, Aarhus University Hospital, DK-8000 Aarhus C, Denmark